CLINICAL TRIAL: NCT04683770
Title: An Observational Study：Prognostic Value of Biomarkers in HR + / HER2 - Advanced Breast Cancer
Brief Title: Prognostic Value of Biomarkers in HR + / HER2 - Advanced Breast Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Jianli Zhao, Attending Doctor, Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Other Study IDs: 2020-KY-063
Record Dates: First submitted 2020-12-19; First posted 2020-12-24 (Actual); Last update posted 2020-12-24 (Actual); Status verified 2020-12

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; biomarker; prognosis
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The object of this study is to detect the gene mutation of tumor tissue or peripheral blood circulation tumor DNA of tumor patients. 10ml of tissue or fresh peripheral blood should be collected as the test sample and stored at room temperature. On the same day, it was sent to the "cell and molecular diagnosis center" of our hospital for DNA isolation and extraction, second-generation sequencing, and detection of related biomarkers. The clinical total exome sequencing (4813 gene) kit developed by Illumina company was used for embryo line detection, and the system detection project used the system detection chip designed by the laboratory.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- HR + / HER2 - advanced breast cancer

SUMMARY:
Our study is aimed to explore a prospective observational clinical study on the efficacy prediction and survival prediction of HR + / HER2 - biomarkers detection in patients with advanced breast cancer. This study is a prospective, observational clinical study. We analyzed the incidence of biomarker mutations in HR + / HER2 - advanced breast cancer (stage IV), and the correlation between biomarkers and therapeutic efficacy, survival, and prognosis.

ELIGIBILITY:
Inclusion Criteria:

1. Adult female patients (aged 18-80 years, including 18 and 80 years) with advanced breast cancer confirmed by pathology or imaging are not suitable for surgical resection or radiotherapy for the purpose of cure;
2. Pathological examination confirmed that ER and/or PR were positive and HER-2 was negative (ER expression: immunohistochemical staining > 1% of tumor cells; PR expression: immunohistochemical staining of tumor cells > 1%; HER-2 negative: immunohistochemical staining of 0,1 +, or fish / CISH negative)
3. No more than four systematic treatments have been used for advanced diseases
4. It is expected that the patients can be followed up at least once after the treatment plan is formulated.
5. The WHO physical status was 0-2 points, and the expected survival time was not less than 3 months;
6. No more than four systematic treatment regimens have been received in the past for advanced diseases
7. There was at least one measurable lesion (short diameter of lymph node ≥ 15mm) in imaging examination within 2 weeks before enrollment, and a conventional CT scan was performed. The diameter of spiral CT scan was more than or equal to 20 mm or more than 10 mm.
8. Prior treatment-related toxicity should be reduced to NCI CTCAE (version 4.03) ≤ 1 degree (except for hair loss or other toxicity judged by the researcher as having no risk to the safety of patients)
9. Within one week before admission, blood routine examination was basically normal: A. white blood cell count (WBC) ≥ 3.0 × 10 ^ 9 / L; B. neutrophil count (ANC) ≥ 1.5 × 10 ^ 9 / L; C. platelet count (PLT) ≥ 100 × 10 ^ 9 / L;
10. Within one week before admission, liver, and kidney function tests were basically normal (based on the normal values of laboratories in each research center): A. total bilirubin (TBIL) ≤ 1.5 × ULN; B. alanine aminotransferase and aspartate aminotransferase (ALT / AST) ≤ 2.5 × ULN (liver metastases ≤ 5xuln); C. serum creatinine ≤ 1.5 × ULN or creatinine clearance rate (CCR) ≥ 60 ml/min；

Exclusion Criteria:

1. The diagnosis of any other malignant tumor within 3 years before enrollment, except for basal cell or squamous cell skin cancer or cervical carcinoma in situ after adequate treatment;
2. Poor compliance or the situation that the researchers think is not suitable to be included in the study;
3. Pregnant or lactating patients;
4. Patients who had received transplantation before;
5. Patients who had previously received stem cell therapy;
6. Patients who have received any immunotherapy that may introduce exogenous DNA and other patients who may introduce exogenous DNA within 4 weeks;
7. Have received more than four systematic treatments for advanced diseases;
8. May interfere with the concomitant diseases or conditions involved in the study, or have any serious medical barriers that may affect the safety of the subjects (e.g., uncontrollable heart disease, hypertension, active or uncontrollable infection, active hepatitis B virus infection);

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Breast Cancer
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2021-07-01 (Estimated); Study Completion 2022-07-01 (Estimated)

PRIMARY OUTCOMES:
Correlation between biomarkers and efficacy of tumor therapy | 1 year
  explore the correlation between biomarkers and the ORR. The biomarkers will be test by nest-generation sequence, which include 520 genes and tumor mutation burden, like ERBB2/TP53/PIK3CA/ERBB4/CCND1 and so on.

SECONDARY OUTCOMES:
overall survival，OS | 2 year
  The time from the beginning of treatment to the death of the patient
Complete remission, CR | 1 year
  all target lesions disappeared, no new lesions appeared, and tumor markers were normal, which lasted for at least 4 weeks
Partial remission, PR | 1 year
  the diameter of target lesions diminished more than 30% and lasted for 4 weeks
Disease stable, SD | 1 year
  the sum of the maximum diameter of the target lesion is smaller than PR, or the increase is not up to PD
Disease progression, PD | 1 year
  the sum of the maximum diameter of the target lesion increased by at least 20%, and its absolute value increased by at least 5 mm, New lesions are also considered as PD
Objective response rate , ORR | 1 year
  according to recist1.1 criteria, the proportion of patients whose best remission is CR or PR in the total number of evaluable patients
Clinical benefit rate, CBR | 1 year
  according to recist1.1 criteria, the proportion of patients with Cr or PR or SD ≥ 24 weeks in the total number of evaluable patients.
Quality of life scale score，QoL | 1 year
  The quality of life score of patients during treatment was analyzed（FACT-B）. Performance Status Rating (PSR) was demonstrated for the FACT-B total score, which is the result of the following subscale scores: SWB (the Social / family Well-Being subscale) , EWB (the Emotional Well-Being subscale), AC (Additional Concerns subscale), PWB (the Physical Well-Being subscale), FWB (the Functional Well-Being subscale)

CONTACTS AND LOCATIONS:
Overall Officials: Jianli Dr. Zhao, doctor, Principal Investigator — Study Principal Investigator
Locations (1):
- Sun Yat Sen Memorial Hospital，Sun Yat sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No